CLINICAL TRIAL: NCT05702359
Title: Acute Effects of Fruit Juice Enriched With Vitamin D3 or n-3 Fatty Acids or Probiotics and the Combination of the Three Ingredients on Glucose Metabolism in Healthy Adults
Brief Title: Acute Effects of Juice Consumption With Biofunctional Compounds and Probiotics on Glucose Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agricultural University of Athens (Other)
Responsible Party: Principal Investigator, Aimilia Papakonstantinou, Assistant Professor, Agricultural University of Athens
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: HRBD 78 12.10.2022
Record Dates: First submitted 2023-01-19; First posted 2023-01-27 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Potential Abnormality of Glucose Tolerance; Appetite Disorders
Keywords: blood glucose; insulin; glycemic index; glycemic load; juices; probiotics; vitamin D3; n-3 fatty acids
MeSH Terms: conditions — Feeding and Eating Disorders; Insulin Resistance | interventions — Glucose; Cholecalciferol; Fatty Acids, Omega-3; Probiotics

STUDY DESIGN:
Intervention Model Description: Crossover assignment
Who Masked: Participant, Investigator
Masking Description: double blind (both the investigator and the participant was not aware of the treatment)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Glucose as reference food (Experimental): Eleven healthy, normal body weight (male: 6, female: 5) adults after a 12hr fast, consumed 50g available carbohydrates from D-glucose, tested two times, in different visits as reference food, along with 300mL water. Fingertip capillary blood glucose samples were collected at baseline and 15, 30, 45, 60, 90, 120, 150, and 180 min after test drink consumption. Salivary insulin samples were collected at baseline, 15, 30, 45, 60, 90, 120, and 180 min after test drink consumption.
  Interventions: Other: Glucose as reference food
- Control juice (Experimental): Eleven healthy, normal body weight (male: 6, female: 5) adults after a 12hr fast, consumed 50g available carbohydrates from control mixed fruit juice (pomegranate, grape, apple and orange), tested once, in random order, along with 300mL water. Fingertip capillary blood glucose samples were collected at baseline and 15, 30, 45, 60, 90, 120, 150, and 180 min after test drink consumption. Salivary insulin samples were collected at baseline, 15, 30, 45, 60, 90, 120, and 180 min after test drink consumption.
  Interventions: Other: Control juice
- Juice containing vitamin D3 (Experimental): Eleven healthy, normal body weight (male: 6, female: 5) adults after a 12hr fast, consumed 50g available carbohydrates from mixed fruit juice enriched with vitamin D3, tested once, in random order, along with 300mL water. Fingertip capillary blood glucose samples were collected at baseline and 15, 30, 45, 60, 90, 120, 150, and 180 min after test drink consumption. Salivary insulin samples were collected at baseline, 15, 30, 45, 60, 90, 120, and 180 min after test drink consumption.
  Interventions: Other: Juice with vitamin D3
- Juice containing n-3 polyunsaturated fatty acids (PUFA) (Experimental): Eleven healthy, normal body weight (male: 6, female: 5) adults after a 12hr fast, consumed 50g available carbohydrates from mixed fruit juice enriched with n-3 PUFA, tested once, in random order, along with 300mL water. Fingertip capillary blood glucose samples were collected at baseline and 15, 30, 45, 60, 90, 120, 150, and 180 min after test drink consumption. Salivary insulin samples were collected at baseline, 15, 30, 45, 60, 90, 120, and 180 min after test drink consumption.
  Interventions: Other: Juice with n-3 fatty acids
- Juice containing probiotics (Experimental): Eleven healthy, normal body weight (male: 6, female: 5) adults after a 12hr fast, consumed 50g available carbohydrates from mixed fruit juice enriched with probiotics, tested once, in random order, along with 300mL water. Fingertip capillary blood glucose samples were collected at baseline and 15, 30, 45, 60, 90, 120, 150, and 180 min after test drink consumption. Salivary insulin samples were collected at baseline, 15, 30, 45, 60, 90, 120, and 180 min after test drink consumption.
  Interventions: Other: Juice with probiotics
- Juice containing probiotics, vitamin D3, and n-3 PUFA (Experimental): Eleven healthy, normal body weight (male: 6, female: 5) adults after a 12hr fast, consumed 50g available carbohydrates from a mixed juice enriched with probiotics, vitamin D3, and n-3 PUFA, tested once, in random order, along with 300mL water. Fingertip capillary blood glucose samples were collected at baseline and 15, 30, 45, 60, 90, 120, 150, and 180 min after test drink consumption. Salivary insulin samples were collected at baseline, 15, 30, 45, 60, 90, 120, and 180 min after test drink consumption.
  Interventions: Other: Juice with probiotics, vitamin D3, and n-3 fatty acids

INTERVENTIONS:
Other: Glucose as reference food — Eleven healthy, normal body weight subjects after 10-14hr fast, consumed 50g glucose diluted in 300mL water, tested two times, in different visits, within 5-10 min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90, 120, 150 and 180 min. Salivary insulin samples were taken at baseline, 15, 30, 45, 60, 90, 120, and 180 min.
  Other Names: reference drink D-Glucose
  Arms: Glucose as reference food
Other: Control juice — Eleven healthy, normal body weight subjects after 10-14hr fast, consumed 50g available carbohydrates from control juice (consisted of pomegranate, grape, apple and orange), tested once, within 5-10 min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90, 120, 150 and 180 min. Salivary insulin samples were taken at baseline, 15, 30, 45, 60, 90, 120, and 180 min.
  Arms: Control juice
Other: Juice with vitamin D3 — Eleven healthy, normal body weight subjects after 10-14hr fast, consumed 50g available carbohydrates from juice (consisted of pomegranate, grape, apple and orange) containing vitamin D3, tested once, within 5-10 min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90, 120, 150 and 180 min. Salivary insulin samples were taken at baseline, 15, 30, 45, 60, 90, 120, and 180 min.
  Other Names: Vitamin D3
  Arms: Juice containing vitamin D3
Other: Juice with n-3 fatty acids — Eleven healthy, normal body weight subjects after 10-14hr fast, consumed 50g available carbohydrates from juice (consisted of pomegranate, grape, apple and orange) containing n-3 fatty acids, tested once, within 5-10 min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90, 120, 150 and 180 min. Salivary insulin samples were taken at baseline, 15, 30, 45, 60, 90, 120, and 180 min.
  Other Names: n-3 fatty acids
  Arms: Juice containing n-3 polyunsaturated fatty acids (PUFA)
Other: Juice with probiotics — Eleven healthy, normal body weight subjects after 10-14hr fast, consumed 50g available carbohydrates from juice (consisted of pomegranate, grape, apple and orange) containing probiotics, tested once, within 5-10 min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90, 120, 150 and 180 min. Salivary insulin samples were taken at baseline, 15, 30, 45, 60, 90, 120, and 180 min.
  Other Names: probiotics
  Arms: Juice containing probiotics
Other: Juice with probiotics, vitamin D3, and n-3 fatty acids — Eleven healthy, normal body weight subjects after 10-14hr fast, consumed 50g available carbohydrates from juice (consisted of pomegranate, grape, apple and orange) containing probiotics, vitamin D3 and n-3 fatty acids, tested once, within 5-10 min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90, 120, 150 and 180 min. Salivary insulin samples were taken at baseline, 15, 30, 45, 60, 90, 120, and 180 min.
  Other Names: probiotics, vitamin D-3, and n-3 fatty acids
  Arms: Juice containing probiotics, vitamin D3, and n-3 PUFA

SUMMARY:
This study investigated the short-term effects of fruit juice enriched with Vitamin D3 or n-3 PUFA or probiotics and the combination of the three ingredients on glucose metabolism.

DETAILED DESCRIPTION:
This study aimed to 1. Determine the glycemic index and glycemic load of mixed fruit juice (pomegranate, grape, apple, and orange) enriched with Vitamin D3 or n-3 PUFA or probiotics, and the combination of the three bio-functional ingredients, compared to regular mixed fruit juice and the reference food (D-glucose), and 2.Examine the short-term effects of the five mixed fruit juices on postprandial blood glucose and salivary insulin responses, blood pressure, and subjective appetite, in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Non-smoking
* Non-diabetic men and women
* Body mass index between 18.5 and 25 kg.m2

Exclusion Criteria:

* Severe chronic disease (e.g. cardiovascular diseases, diabetes mellitus, kidney or liver conditions, endocrine conditions)
* Gastrointestinal disorders
* Pregnancy
* Lactation
* Competitive sports
* Alcohol abuse
* Drug dependency

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Capillary blood glucose responses | 3 hours
  Clinically useful change in blood glucose, defined as the restoration of glucose within normal limits during the 3hr glucose tolerance test

SECONDARY OUTCOMES:
Salivary insulin responses | 3 hours
  Clinically useful change in salivary insulin, defined as the restoration of insulin within normal limits during the 3hr glucose torelance test
Subjective appetite rating | 3 hours
  Useful change in subjective appetite using visual analogue scales (VAS). Participants rated their hunger, desire to eat, perceived fullness, thirst, preoccupation with food, pleasure of eating the consumed test food, and thirst, after eating on a horizontal line VAS, with a line length of 10 cm, a line width of 3 desktop publishing points, was black, had flat line endpoints, had an ascending numerical order of scale endpoints [i.e., "0" and "10", for example neither hungry (0 mm), full (100 mm) or have desire for food in the middle (50 mm)], and used "0" and "10" as numerical anchors below the left and right endpoints, respectively.
Blood pressure | 3 hours
  Useful change in systolic and diastolic blood pressure before and 3hr after consumption of the juices.

CONTACTS AND LOCATIONS:
Overall Officials: Emilia Papakonstantinou, PhD, Principal Investigator — Agricultural University of Athens
Locations (1):
- Agricultural University of Athens, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No